CLINICAL TRIAL: NCT01295801
Title: The Effects and Mechanism of Vitamin B6 on Relieving Linezolid-associated Cytopenias
Brief Title: Vitamin B6 on Relieving Linezolid-associated Cytopenias
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Lixin Xie, Pneumology Department of Chinese PLA General Hospital
Other Study IDs: 301PLAGH-20101027001
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2010-10

CONDITIONS: Cytopenias; Erythropenia (Diagnosis)
Keywords: Linezolid; Vitamin B6; Linezolid-associated cytopenias
MeSH Terms: conditions — Cytopenia; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Linezolid+vitamin B6
- Linezolid

SUMMARY:
Linezolid is the first approved synthetic oxazolidinone that is active against multidrug-resistant Gram-positive pathogens. Because of its significant efficacy, linezolid is widely used in clinical treatment. However, the side effects of linezolid commonly lead to anemia and thrombocytopenia. This hematological toxic effects limit its prolonged used. The investigators have found that Vitamin B6 application, as a preventive, auxiliary therapy, can relieve anemia and thrombocytopenia. The present study was designed to verify the effects of Vitamin B6 in the prevention of linezolid-associated cytopenias and investigate its mechanism.

DETAILED DESCRIPTION:
Infected patients receiving linezolid therapy are divided into two groups, i.e. the linezolid group and the linezolid + vitamin B6 group, the line of division being whether vitamin B6 is to be applied or not in the course of treatment. The purpose is to evaluate the role that vitamin B6 plays, during the process of linezolid therapy, in the relief of erythropenia and cytopenias.

ELIGIBILITY:
Inclusion Criteria:

* Use of linezolid is not less than 3 days

Exclusion Criteria:

* Serious adverse reactions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Use of linezolid
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-07 (Estimated); Study Completion 2011-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Xie Lixin, Doctor, Study Director — Pneumology Department of chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Deng J, Su LX, Liang ZX, Liang LL, Yan P, Jia YH, Zhang XG, Feng D, Xie LX. Effects of vitamin b6 therapy for sepsis patients with linezolid-associated cytopenias: a retrospective study. Curr Ther Res Clin Exp. 2013 Jun;74:26-32. doi: 10.1016/j.curtheres.2012.12.002. PMID 24385027